CLINICAL TRIAL: NCT05138614
Title: Supporting Treatment Access and Recovery in Co-Occurring Opioid Use and Mental Health Disorders
Brief Title: Supporting Treatment Access and Recovery in COD
Acronym: STAR-COD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Massachusetts, Lowell (Other); Cornell University (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, David Smelson, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: H00023911; 1R01MH128904 (NIH)
Record Dates: First submitted 2021-10-22; First posted 2021-12-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use Disorder; Mental Health Disorder
Keywords: opioid use disorder; mental health
MeSH Terms: conditions — Opioid-Related Disorders; Mental Disorders; Psychological Well-Being | interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: MISSION is a time-limited, cross disciplinary, team-based wraparound approach that provides 6 months of psychosocial treatment combined with assertive outreach, empowering clients to access and engage in care and community services to promote recovery. The MISSION treatment curriculum integrates 3 evidence-based practices along with MOUD: 1) Critical Time Intervention (CTI), a time-limited form of assertive community treatment; 2) Dual Recovery Therapy (DRT), which is integrated mental health and substance use group therapy; and 3) Peer Support (PS), offering support for people in recovery by people in recovery
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Full MISSION (Experimental): CTI + DRT + PS + MOUD
  Interventions: Other: Medication for Opioid Use Disorder; Behavioral: MISSION Critical Time Intervention; Behavioral: MISSION Peer Support; Behavioral: MISSION Dual Recovery Therapy
- CTI & DRT (Experimental): CTI + DRT + MOUD
  Interventions: Other: Medication for Opioid Use Disorder; Behavioral: MISSION Critical Time Intervention; Behavioral: MISSION Dual Recovery Therapy
- CTI & PS (Experimental): CTI + PS + MOUD
  Interventions: Other: Medication for Opioid Use Disorder; Behavioral: MISSION Critical Time Intervention; Behavioral: MISSION Peer Support
- DRT & PS (Experimental): DRT + PS + MOUD
  Interventions: Other: Medication for Opioid Use Disorder; Behavioral: MISSION Peer Support; Behavioral: MISSION Dual Recovery Therapy
- MOUD only (Other): MOUD
  Interventions: Other: Medication for Opioid Use Disorder

INTERVENTIONS:
Other: Medication for Opioid Use Disorder — medication management
  Other Names: MOUD
Behavioral: MISSION Critical Time Intervention — offering intensive community-based services that decrease in intensity over time
  Other Names: CTI
  Arms: CTI & DRT; CTI & PS; Full MISSION
Behavioral: MISSION Peer Support — including 11 recovery-oriented sessions from someone with lived experience of co-occurring disorders
  Other Names: PS
  Arms: CTI & PS; DRT & PS; Full MISSION
Behavioral: MISSION Dual Recovery Therapy — comprised of 13 structured co-occurring disorders treatment sessions
  Other Names: DRT
  Arms: CTI & DRT; DRT & PS; Full MISSION

SUMMARY:
This 4-year study will randomize 1,000 people with co-occurring opioid use and mental health disorders (COD) at medication for opioid use disorder (MOUD) clinics to evaluate the effectiveness of MISSION, a multi-component team approach, or its components with MOUD versus MOUD alone, as well as the incremental benefits of MISSION or its components for improving outcomes. We expect that individuals receiving MISSION or its parts + MOUD will show greater improvement over MOUD alone on: engagement, substance use, and mental health.

DETAILED DESCRIPTION:
This is a 5-arm randomized control trial with a fractional factorial design among 1,000 patients across Massachusetts. Patients will be randomized to: 1) MOUD alone; 2) full MISSION (CTI & DRT & PS) + MOUD; 3) CTI & DRT + MOUD; 4) PS & DRT + MOUD; or 5) CTI & PS + MOUD (Arms 3-5 are the 3 combinations of 2 MISSION parts). MISSION is a time-limited, cross disciplinary, team-based wraparound approach that provides 6 months of psychosocial treatment combined with assertive outreach, empowering clients to access and engage in care and community services to promote recovery. The MISSION treatment curriculum integrates 3 evidence-based practices along with MOUD: 1) Critical Time Intervention (CTI), a time-limited form of assertive community treatment; 2) Dual Recovery Therapy (DRT), which is integrated mental health and substance use group therapy; and 3) Peer Support (PS), offering support for people in recovery by people in recovery. Participants will receive 6 months of treatment and be followed for 1-year.

Study aims include:

Aim 1: To evaluate the effectiveness of MISSION or its bundled parts with MOUD versus MOUD alone, as well as the incremental benefits of MISSION and its parts + MOUD to improve outcomes 1a-c for CODs.

Hypothesis 1.1: Individuals receiving MISSION or its parts + MOUD will show greater improvement over MOUD alone on: 1a. Engagement (measured by total days in treatment, percentage of days receiving MOUD, and total number of outreach and linkages sessions); 1b. Opioid use and other substance use (measured by self-report days of use and drug screens); and 1c. Mental health (measured by self-report mental health symptoms).

Hypothesis 1.2: MISSION + MOUD will outperform its parts + MOUD but at least one of the three combinations + MOUD will be at least 75% as effective compared to the full MISSION protocol on outcomes 1a-c.

Aim 2: To examine mechanisms of action of MISSION in CODs. Hypothesis 2.1: The effects of MISSION and its bundled parts on health outcomes (mental health, opioid and other substance use) are mediated by treatment participation and other measures (e.g., recovery capital, psychosocial supports, and quality of life). Hypothesis 2.2: The effects of MISSION and its parts on health outcomes are moderated by key patient characteristics (e.g., demographics, severity of COD, and MOUD type).

Aim 3: To conduct a comprehensive economic evaluation of MISSION or its bundled parts and MOUD.

Estimate cost of full MISSION or its bundled parts compared to MOUD alone, and to evaluate cost-effectiveness and return on investment from multiple perspectives, including patient, clinic, healthcare, taxpayer, and societal.

Exploratory Aim: 4. To construct a predictive model that can match optimum combined use of MISSION parts with specific patient's needs for greater improvements in health outcomes, which will inform a future randomized controlled trial on cost-effective patient-level precision intervention assignment.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years-old and older;
* Are fluent in English or Spanish;
* Have OUD who (a) are newly admitted into the program with OUD; or (b) who have been active in the program for the treatment of OUD with medications like buprenorphine or naltrexone, but experienced a recent relapse with any substance (e.g., alcohol, cocaine, opioids, or benzodiazepines). This second group is necessary to include because patients who may have been stable for a long period of time may have a relapse and need intensive treatment to help them regain their abstinence and facilitate the path towards recovery. Thus, by taking those newly enrolled and those who were stable on MOUD but had a recent relapse, the second group is clinically similar to the first group and the intervention will be meaningful.;
* Able to provide consent;
* Potentially have a concurrent substance use disorder in addition to opioids; and
* Have a co-occurring mental health disorder (COD) including depression, anxiety, trauma-related disorders, bipolar, and/or schizophrenia, and those who are stable on buprenorphine or naltrexone but have recurrence or worsening at any time of symptoms of any co-occurring mental health disorder (COD) including depression, anxiety, trauma-related disorders, bipolar, and/or schizophrenia, even if the patient has not relapsed. Instability is defined in two ways in the study: (a) a substance use relapse; and (b) recurrence to symptom exacerbation in regard to a subject's mental health disorder(s). If subjects do not meet criteria for "a" (i.e., not having a substance use relapse), but they do meet criteria for "b" (i.e., they do in fact have worsening of mental health symptoms), they are then defined as unstable, and will meet study inclusion criteria.

Exclusion Criteria:

* Are not fluent in English or Spanish;
* Are acutely psychotic, acutely suicidal with a plan, or homicidal;
* Are incompetent and unable to provide informed consent; and
* Have concurrent severe alcohol use disorder or high dose benzodiazepine needing detoxification. This exclusion factor is based on DSM-5 criteria, and those who are currently drinking or with a history of severe alcohol withdrawal (i.e., alcohol related seizures, and delirium tremens) will also be excluded. High dose benzodiazepine is defined as using Lorazepam equivalent of > 10 mg/day; Diazepam > 100 mg/day; Clonazepam 5 mg/ day; Alprazolam 5 mg/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Engagement in treatment | 6 months
  Measured by total days in treatment
Engagement in medication for opioid use disorder (MOUD) | 6 months
  Measured by percentage of days receiving MOUD
Engagement in outreach and linkage sessions | 6 months
  Measured by total number of outreach and linkage sessions
Self-report opioid use and other substance use | Baseline
  Measured by self-report days of use
Self-report opioid use and other substance use | 3 months
  Measured by self-report days of use
Self-report opioid use and other substance use | 6 months
  Measured by self-report days of use
Self-report opioid use and other substance use | 9 months
  Measured by self-report days of use
Self-report opioid use and other substance use | 12 months
  Measured by self-report days of use
Opioid use and other substance use (drug screen) | 3 months
  Measured by positive drug screens
Opioid use and other substance use (drug screen) | 6 months
  Measured by positive drug screens
Mental health functioning | Baseline
  Measured by self-report mental health symptoms on Behavior and Symptom Identification Scale (BASIS-24)
Mental health functioning | 3 months
  Measured by self-report mental health symptoms on BASIS-24
Mental health functioning | 6 months
  Measured by self-report mental health symptoms on BASIS-24
Mental health functioning | 9 months
  Measured by self-report mental health symptoms on BASIS-24
Mental health functioning | 12 months
  Measured by self-report mental health symptoms on BASIS-24
PTSD symptoms | Baseline
  Measured by self-report PTSD symptoms on Patient Checklist (PCL-5)
PTSD symptoms | 3 months
  Measured by self-report PTSD symptoms on Patient Checklist (PCL-5)
PTSD symptoms | 6 months
  Measured by self-report PTSD symptoms on Patient Checklist (PCL-5)
PTSD symptoms | 9 months
  Measured by self-report PTSD symptoms on Patient Checklist (PCL-5)
PTSD symptoms | 12 months
  Measured by self-report PTSD symptoms on Patient Checklist (PCL-5)
Mental health impairment | Baseline
  Measured by self-report on World Health Organization Disability Assessment (WHODAS 2.0)
Mental health impairment | 3 months
  Measured by self-report on WHODAS 2.0
Mental health impairment | 6 months
  Measured by self-report on WHODAS 2.0
Mental health impairment | 9 months
  Measured by self-report on WHODAS 2.0
Mental health impairment | 12 months
  Measured by self-report on WHODAS 2.0
Psychiatric severity | Baseline
  Measured by Structured Clinical Interview for DSM-5 (SCID-RV)
Health functioning | Baseline
  Measured by the World Health Organization Quality of Life Scale Brief Version (WHOQOL-BREF)
Health functioning | 3 months
  Measured by the WHOQOL-BREF
Health functioning | 6 months
  Measured by the WHOQOL-BREF
Health functioning | 9 months
  Measured by the WHOQOL-BREF
Health functioning | 12 months
  Measured by the WHOQOL-BREF
Motivation for treatment | Baseline
  Measured by Stages of Change, Readiness, and Treatment Eagerness Scale (SOCRATES)
Motivation for treatment | 3 months
  Measured by SOCRATES
Motivation for treatment | 6 months
  Measured by SOCRATES
Motivation for treatment | 9 months
  Measured by SOCRATES
Motivation for treatment | 12 months
  Measured by SOCRATES
Suicide Severity | Baseline
  Measured by Columbia- Suicide Severity Rating Scale (C-SSRS)
Suicide Severity | 3 months
  Measured by C-SSRS
Suicide Severity | 6 months
  Measured by C-SSRS
Suicide Severity | 9 months
  Measured by C-SSRS
Suicide Severity | 12 months
  Measured by C-SSRS
Therapeutic alliance | Baseline
  Measured by Working Alliance Inventory
Therapeutic alliance | 3 months
  Measured by Working Alliance Inventory
Therapeutic alliance | 6 months
  Measured by Working Alliance Inventory
Therapeutic alliance | 9 months
  Measured by Working Alliance Inventory
Therapeutic alliance | 12 months
  Measured by Working Alliance Inventory
Recovery Capital | Baseline
  Measured by Assessment of Recovery Capital
Recovery Capital | 3 months
  Measured by Assessment of Recovery Capital
Recovery Capital | 6 months
  Measured by Assessment of Recovery Capital
Recovery Capital | 9 months
  Measured by Assessment of Recovery Capital
Recovery Capital | 12 months
  Measured by Assessment of Recovery Capital
Chronic pain | Baseline
  Measured by Chronic Pain assessment
Chronic pain | 3 months
  Measured by Chronic Pain assessment
Chronic pain | 6 months
  Measured by Chronic Pain assessment
Chronic pain | 9 months
  Measured by Chronic Pain assessment
Chronic pain | 12 months
  Measured by Chronic Pain assessment
Medication Adherence | 3 months
  Measured by Medication Adherence Rating Scale
Medication Adherence | 6 months
  Measured by Medication Adherence Rating Scale

SECONDARY OUTCOMES:
Mortality | 6 months
  Data extracted from medical records
Quality Adjusted Life Years (QALYs): health | Baseline
  Measured by self-report on the 5-level EQ-5D (EQ-5D-5L). Scores range from 0 (worst imaginable health) to 100 (best imaginable health).
Quality Adjusted Life Years (QALYs): health | 3 months
  Measured by self-report on the 5-level EQ-5D (EQ-5D-5L). Scores range from 0 (worst imaginable health) to 100 (best imaginable health).
Quality Adjusted Life Years (QALYs): health | 6 months
  Measured by self-report on the 5-level EQ-5D (EQ-5D-5L). Scores range from 0 (worst imaginable health) to 100 (best imaginable health).
Quality Adjusted Life Years (QALYs): health | 9 months
  Measured by self-report on the 5-level EQ-5D (EQ-5D-5L). Scores range from 0 (worst imaginable health) to 100 (best imaginable health).
Quality Adjusted Life Years (QALYs): health | 12 months
  Measured by self-report on the 5-level EQ-5D (EQ-5D-5L). Scores range from 0 (worst imaginable health) to 100 (best imaginable health).
Quality Adjusted Life Years (QALYs): quality of life | Baseline
  Measured by self-report on Patient Reported Outcomes - Preference (PROPr). Scores range from 0 to 100 with higher scores indicating worse quality of life.
Quality Adjusted Life Years (QALYs): quality of life | 3 months
  Measured by self-report on Patient Reported Outcomes - Preference (PROPr). Scores range from 0 to 100 with higher scores indicating worse quality of life.
Quality Adjusted Life Years (QALYs): quality of life | 6 months
  Measured by self-report on Patient Reported Outcomes - Preference (PROPr). Scores range from 0 to 100 with higher scores indicating worse quality of life.
Quality Adjusted Life Years (QALYs): quality of life | 9 months
  Measured by self-report on Patient Reported Outcomes - Preference (PROPr). Scores range from 0 to 100 with higher scores indicating worse quality of life.
Quality Adjusted Life Years (QALYs): quality of life | 12 months
  Measured by self-report on Patient Reported Outcomes - Preference (PROPr). Scores range from 0 to 100 with higher scores indicating worse quality of life.

OTHER OUTCOMES:
Economic impact of full MISSION | 6 months
  Cost of full MISSION and MOUD measured by Patient-Reported Outcomes Measurement Information System-Preference (PROPr)
Economic impact of CTI & PS | 6 months
  Cost of MISSION CTI, PS, and MOUD measured by PROPr
Economic impact of CTI & DRT | 6 months
  Cost of MISSION CTI, DRT, and MOUD measured by PROPr
Economic impact of PS & DRT | 6 months
  Cost of MISSION PS, DRT, and MOUD measured by PROPr
Economic impact of MOUD alone | 6 months
  Cost of MOUD alone measured by PROPr

CONTACTS AND LOCATIONS:
Overall Officials: David Smelson, PsyD, Principal Investigator — University of Massachusetts, Worcester
Locations (5):
- United States (5):
  - Behavioral Health Network, Holyoke, Massachusetts
  - Behavioral Health Network, Orange, Massachusetts
  - Behavioral Health Network, Springfield, Massachusetts
  - UMass Chan Road to Care Clinic, Worcester, Massachusetts
  - SaVida Health, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Consistent with the NIH HEAL Initiative, Underlying Primary Data collected from participants in this project will be made readily available to the public through twice-yearly submissions to the NIMH Data Archive (NDA). In consultation with the University of Massachusetts Medical School's institutional review board (IRB), project consent forms will include relevant information for participants to be made aware that their de-identified data will be available to other investigators as a part of the HEAL Initiative Public Access and Data Sharing Policy.
Supporting Information: Study Protocol
Time Frame: Data will be available upon publication (via an NDA Study) or 1-2 years after the grant end date (August 2026), until 2032 (expiration of NDA Certificate of Confidentiality)
Access Criteria: Data will be shared with authorized NDA users.
URL: https://nda.nih.gov/